CLINICAL TRIAL: NCT02482584
Title: DiaBOSA: Impact of CPAP Treatment on Arterial Stiffness in Patients With Type 2 Diabetes and Newly Diagnosed Obstructive Sleep Apnoea
Brief Title: Impact of CPAP Treatment on Arterial Stiffness in Patients With T2DM and Newly Diagnosed Obstructive Sleep Apnoea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DiaBOSA
Record Dates: First submitted 2015-03-31; First posted 2015-06-26 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2016-11

CONDITIONS: Diabetes; Obstructive Sleep Apnea
MeSH Terms: conditions — Diabetes Mellitus; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPAP treatment (Active Comparator): Continuous Positive Airway Pressure (CPAP) treatment during three month.
  Interventions: Device: CPAP
- Control group (Other): Control group
  Interventions: Other: Control

INTERVENTIONS:
Device: CPAP — CPAP intervention
  Arms: CPAP treatment
Other: Control — Control
  Arms: Control group

SUMMARY:
The purpose of the trial is to investigate the effects of three months' treatment with a CPAP-device versus control group on change in arterial stiffness in type 2 diabetes (T2D) patients with newly detected Obstructive Sleep Apnoea (OSA).

DETAILED DESCRIPTION:
Background: Obstructive sleep apnoea (OSA) is a common disorder characterised by recurrent episodes of apnoea or hypopnoea during sleep. OSA is associated with excessive daytime sleepiness and linked to increased cardiovascular morbidity and mortality. OSA can be alleviated with Continuous Positive Airway Pressure (CPAP) treatment.

Cardiovascular disease is the major cause of decreased life expectancy, morbidity and reduced quality of life in patients with type 2 diabetes (T2D). Increased stiffness of the aorta has been associated with increased cardiovascular morbidity and mortality in diabetic patients.

Previous studies have reported a much higher frequency of OSA in patients with obesity and T2D compared with non-diabetic subjects, and found that OSA was associated with arterial stiffness. However, whether CPAP treatment improves arterial stiffness and insulin sensitivity in T2D patients remain to be elucidated.

Objective: To investigate the effects of three months' treatment with a CPAP-device versus sham CPAP on change in arterial stiffness in T2D patients with newly detected OSA.

Design: Randomised, controlled, multicentre study of intervention with CPAP treatment versus control group. The treatment period is three months with a subsequent 9 months open extension.

Patient population: 70 patients with T2D and newly diagnosed OSA recruited from Department of Cardiology, Nephrology and Endocrinology, Nordsjællands Hospital, Department of Endocrinology, Gentofte University Hospital, Department of Endocrinology and Internal Medicine, Aarhus University Hospital Nørrebrogade and Department of Internal Medicine, Silkeborg Sygehus.

Intervention: CPAP treatment versus control group.

Endpoints:

Primary endpoint: Change in arterial stiffness measured by office carotid-femoral pulse wave velocity (cf-PWV) from start to end of 12 weeks intervention.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (WHO criteria)
* Obstructive sleep apnea defined as apnoea-hypopnoea index (AHI) > 15 diagnosed with ApneaLink+® measured within three months or less prior to visit 0.
* Signed informed content.

Exclusion Criteria:

* Contraindications to CPAP treatment.
* Treatment with CPAP within the last 6 months prior to visit 1.
* Works in a transportation-related industry
* C-peptide < 300 pmol/l - measured less than 6 months prior to visit 0
* HbA1c:< 7% or >10% - both exclusive - at visit 0
* Changes in antidiabetic treatment during the last four weeks prior to visit 0.
* Unstable bodyweight, i.e. >5% change during the last three months prior to visit 0.
* Other sleep breathing disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-02 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Change in arterial stiffness measured by office carotid-femoral pulse wave velocity (cf-PWV) from start to end of 12 weeks intervention | three month

SECONDARY OUTCOMES:
Change from start to end of 13 weeks intervention in insulin sensitivity measured by hyperinsulinemic euglycemic clamp | three month

CONTACTS AND LOCATIONS:
Overall Officials: Esben Laugesen, MD, Principal Investigator — Aarhus Universitets Hospital
Locations (1):
- Nordsjællands hospital, Hillerød, Denmark

REFERENCES:
- [Derived] Hvelplund Kristiansen M, Banghoj AM, Laugesen E, Tarnow L. Arterial stiffness in people with Type 2 diabetes and obstructive sleep apnoea. Diabet Med. 2018 Oct;35(10):1391-1398. doi: 10.1111/dme.13666. Epub 2018 May 24. PMID 29763980